CLINICAL TRIAL: NCT06405659
Title: Immediate Fever During Anaesthesia Recovery After Surgical Procedure With Scoliosis: A Case Report and Literature Review
Brief Title: Immediate Fever During Anaesthesia Recovery After Surgical Procedure With Scoliosis
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: YJLW2019001
Record Dates: First submitted 2024-04-24; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Fever; Scoliosis; Surgical Trauma; Hypothermia; General Anaesthesia
MeSH Terms: conditions — Fever; Scoliosis; Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: correction for pedicle fixation — The patient was diagnosed with idiopathic scoliosis and underwent a posterior idiopathic scoliosis procedure and correction for pedicle fixation.

SUMMARY:
Fever is a common clinical symptom in patients with postoperative scoliosis. However, there are rare reports of immediately fevers occurring following operative procedures.

DETAILED DESCRIPTION:
Postoperative fever is a common clinical symptom in patients following spinal surgery, with an incidence of 13.2%, and 64.5% of patients with neuromuscular scoliosis were observed to develop postoperative fevers. The most frequently observed cause of fever is surgical trauma, which is associated with inflammatory responses to surgery, and such fevers typically resolve within 2-3 days. This self-limited cause of postoperative fever is non-pathological,4 and the severity and duration of such fevers depend on the duration, scope, and type of surgery, and whether a mesh graft was inserted. The aetiology of immediate postoperative fever for patients following hip prosthesis implantation is unknown, and it is inexpedient to initiate antibiotic treatment or to increase the prophylactic antibiotic dosage. However, there are rare reports of chills and fevers occurring immediately following spinal surgery, to the best of our knowledge, there have been no reports on the mechanism of immediate postoperative fever following spinal surgery.

Based on this evidence and on observation, when patients experience postoperative fevers, nearly all surgeons seek to exclude infection as a cause. The case presented in this paper is that of a 15-year-old female with idiopathic scoliosis who underwent posterior idiopathic scoliosis incision and correction for pedicle fixation. The clinical symptoms of interest, including chills, a high fever, an increased heart rate and increased blood pressure, were observed immediately during the course of anaesthesia resuscitation. In this report, risk factors, treatment and prevention are assessed based on the case evidence.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A 15-year-old female with a 1-year history of scoliosis was admitted to the hospital after a health examination.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
surgical complication | up to 3 years, after surgical procedure
  Complications related to the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yiyue Zhong, Ph.D., Principal Investigator — Affiliated Hospital of Guangdong Medical University
Locations (1):
- The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The raw data for this case and related of cases can be obtained from corresponding authors YYZ by e-mail.

REFERENCES:
- [Background] Yousef MAA, Rosenfeld S. Evaluation of postoperative fever after surgical correction of neuromuscular scoliosis: implication on management. Eur Spine J. 2018 Aug;27(8):1690-1697. doi: 10.1007/s00586-017-5456-1. Epub 2018 Jan 9. PMID 29318413
- [Background] Petretta R, McConkey M, Slobogean GP, Handel J, Broekhuyse HM. Incidence, risk factors, and diagnostic evaluation of postoperative fever in an orthopaedic trauma population. J Orthop Trauma. 2013 Oct;27(10):558-62. doi: 10.1097/BOT.0b013e31828af4df. PMID 23412504
- [Background] Blumstein GW, Andras LM, Seehausen DA, Harris L, Ross PA, Skaggs DL. Fever is common postoperatively following posterior spinal fusion: infection is an uncommon cause. J Pediatr. 2015 Mar;166(3):751-5. doi: 10.1016/j.jpeds.2014.11.033. Epub 2015 Jan 6. PMID 25575423
- [Background] Clark JA, Bar-Yosef S, Anderson A, Newman MF, Landolfo K, Grocott HP. Postoperative hyperthermia following off-pump versus on-pump coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2005 Aug;19(4):426-9. doi: 10.1053/j.jvca.2005.01.042. PMID 16085244
- [Background] Sharp NE, Alemayehu H, Desai A, Holcomb GW 3rd, St Peter SD. Fever after redo Nissen fundoplication with hiatal hernia repair. J Surg Res. 2014 Aug;190(2):594-7. doi: 10.1016/j.jss.2014.05.021. Epub 2014 May 14. PMID 24948540
- [Background] Zhao Z, Ma X, Ma J, Sun X, Li F, Lv J. A Systematic Review and Meta-analysis of the Topical Administration of Fibrin Sealant in Total Hip Arthroplasty. Sci Rep. 2018 Jan 8;8(1):78. doi: 10.1038/s41598-017-16779-3. PMID 29311570
- [Background] Badillo AT, Sarani B, Evans SR. Optimizing the use of blood cultures in the febrile postoperative patient. J Am Coll Surg. 2002 Apr;194(4):477-87; quiz 554-6. doi: 10.1016/s1072-7515(02)01115-8. No abstract available. PMID 11949753
- [Background] de la Torre SH, Mandel L, Goff BA. Evaluation of postoperative fever: usefulness and cost-effectiveness of routine workup. Am J Obstet Gynecol. 2003 Jun;188(6):1642-7. doi: 10.1067/mob.2003.397. PMID 12825005
- [Background] Walid MS, Sahiner G, Robinson C, Robinson JS 3rd, Ajjan M, Robinson JS Jr. Postoperative fever discharge guidelines increase hospital charges associated with spine surgery. Neurosurgery. 2011 Apr;68(4):945-9; discussion 949. doi: 10.1227/NEU.0b013e318209c80a. PMID 21242842
- [Background] Krishnan SS, Nigam P, Bachh O, Vasudevan MC. Quad Fever: Treatment through Lowering of Ambient Temperature. Indian J Crit Care Med. 2018 Jan;22(1):43-45. doi: 10.4103/ijccm.IJCCM_295_17. PMID 29422733
- [Background] Abeysinghe P, Ekanayake H, Ranasinghe J. Transfusion related acute lung injury (TRALI)-a case report. Vox Sanguinis 2017; 112: 273.
- [Background] Pile JC. Evaluating postoperative fever: a focused approach. Cleve Clin J Med. 2006 Mar;73 Suppl 1:S62-6. doi: 10.3949/ccjm.73.suppl_1.s62. PMID 16570551
- [Background] Sloan TB, Myers G, Janik DJ, Burger EM, Patel VV, Jameson LC. Intraoperative autologous transfusion of hemolyzed blood. Anesth Analg. 2009 Jul;109(1):38-42. doi: 10.1213/ane.0b013e3181a335e4. PMID 19535693
- [Background] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Background] MacLennan DH, Phillips MS. Malignant hyperthermia. Science. 1992 May 8;256(5058):789-94. doi: 10.1126/science.1589759.
- [Background] Anetseder M, Hager M, Muller CR, Roewer N. Diagnosis of susceptibility to malignant hyperthermia by use of a metabolic test. Lancet. 2002 May 4;359(9317):1579-80. doi: 10.1016/S0140-6736(02)08506-9. PMID 12047971
- [Background] Gray RM. Anesthesia-induced rhabdomyolysis or malignant hyperthermia: is defining the crisis important? Paediatr Anaesth. 2017 May;27(5):490-493. doi: 10.1111/pan.13130. Epub 2017 Mar 17. PMID 28306187
- [Background] Sadrolsadat SH, Mahdavi AR, Moharari RS, Khajavi MR, Khashayar P, Najafi A, Amirjamshidi A. A prospective randomized trial comparing the technique of spinal and general anesthesia for lumbar disk surgery: a study of 100 cases. Surg Neurol. 2009 Jan;71(1):60-5; discussion 65. doi: 10.1016/j.surneu.2008.08.003. PMID 19084683
- [Background] Ren Z, He S, Li J, Wang Y, Lai J, Sun Z, Feng H, Wang J. Comparison of the Safety and Effectiveness of Percutaneous Endoscopic Lumbar Discectomy for Treating Lumbar Disc Herniation Under Epidural Anesthesia and General Anesthesia. Neurospine. 2020 Mar;17(1):254-259. doi: 10.14245/ns.1938366.183. Epub 2020 Feb 1. PMID 32054145
- [Background] Carr DB, Bergland R, Hamilton A, Blume H, Kasting N, Arnold M, Martin JB, Rosenblatt M. Endotoxin-stimulated opioid peptide secretion: two secretory pools and feedback control in vivo. Science. 1982 Aug 27;217(4562):845-8. doi: 10.1126/science.6285473.
- [Background] Ezhevskaya AA, Mlyavykh SG, Anderson DG. Effects of continuous epidural anesthesia and postoperative epidural analgesia on pain management and stress response in patients undergoing major spinal surgery. Spine (Phila Pa 1976). 2013 Jul 1;38(15):1324-30. doi: 10.1097/BRS.0b013e318290ff26. PMID 23514874
- [Background] Lenhardt R. The effect of anesthesia on body temperature control. Front Biosci (Schol Ed). 2010 Jun 1;2(3):1145-54. doi: 10.2741/s123. PMID 20515846
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] Feketa VV, Zhang Y, Cao Z, Balasubramanian A, Flores CM, Player MR, Marrelli SP. Transient receptor potential melastatin 8 channel inhibition potentiates the hypothermic response to transient receptor potential vanilloid 1 activation in the conscious mouse. Crit Care Med. 2014 May;42(5):e355-63. doi: 10.1097/CCM.0000000000000229. PMID 24595220
- [Background] Tan CL, Cooke EK, Leib DE, Lin YC, Daly GE, Zimmerman CA, Knight ZA. Warm-Sensitive Neurons that Control Body Temperature. Cell. 2016 Sep 22;167(1):47-59.e15. doi: 10.1016/j.cell.2016.08.028. Epub 2016 Sep 8. PMID 27616062
- [Background] Cheon YM, Yoon H. [The Effects of 30-Minutes of Pre-Warming on Core Body Temperature, Systolic Blood Pressure, Heart Rate, Postoperative Shivering, and Inflammation Response in Elderly Patients with Total Hip Replacement under Spinal Anesthesia: A Randomized Double-blind Controlled Trial]. J Korean Acad Nurs. 2017 Aug;47(4):456-466. doi: 10.4040/jkan.2017.47.4.456. Korean. PMID 28894068
- [Background] Cobb B, Cho Y, Hilton G, Ting V, Carvalho B. Active Warming Utilizing Combined IV Fluid and Forced-Air Warming Decreases Hypothermia and Improves Maternal Comfort During Cesarean Delivery: A Randomized Control Trial. Anesth Analg. 2016 May;122(5):1490-7. doi: 10.1213/ANE.0000000000001181. PMID 26895002
- [Background] Steelman VM, Chae S, Duff J, Anderson MJ, Zaidi A. Warming of Irrigation Fluids for Prevention of Perioperative Hypothermia During Arthroscopy: A Systematic Review and Meta-analysis. Arthroscopy. 2018 Mar;34(3):930-942.e2. doi: 10.1016/j.arthro.2017.09.024. Epub 2017 Dec 6. PMID 29217304
- [Background] Aarnes TK, Bednarski RM, Lerche P, Hubbell JA. Effect of pre-warming on perioperative hypothermia and anesthetic recovery in small breed dogs undergoing ovariohysterectomy. Can Vet J. 2017 Feb;58(2):175-179. PMID 28216687
- [Background] Santa Maria PL, Santa Maria C, Eisenried A, Velasquez N, Kannard BT, Ramani A, Kahn DM, Wheeler AJ, Brock-Utne JG. A novel thermal compression device for perioperative warming: a randomized trial for feasibility and efficacy. BMC Anesthesiol. 2017 Aug 11;17(1):102. doi: 10.1186/s12871-017-0395-2. PMID 28800725
- [Background] Torossian A, Van Gerven E, Geertsen K, Horn B, Van de Velde M, Raeder J. Active perioperative patient warming using a self-warming blanket (BARRIER EasyWarm) is superior to passive thermal insulation: a multinational, multicenter, randomized trial. J Clin Anesth. 2016 Nov;34:547-54. doi: 10.1016/j.jclinane.2016.06.030. Epub 2016 Jul 17. PMID 27687449
- [Background] Zeba S, Surbatovic M, Marjanovic M, Jevdjic J, Hajdukovic Z, Karkalic R, Jovanovic D, Radakovic S. Efficacy of external warming in attenuation of hypothermia in surgical patients. Vojnosanit Pregl. 2016 Jun;73(6):566-71. doi: 10.2298/vsp150330032z. PMID 27498449
- [Background] Lee WP, Wu PY, Shih WM, Lee MY, Ho LH. The effectiveness of the newly designed thermal gown on hypothermic patients after spinal surgery. J Clin Nurs. 2015 Oct;24(19-20):2779-87. doi: 10.1111/jocn.12873. Epub 2015 Jul 5. PMID 26147373
- [Background] Fujita T, Okada N, Kanamori J, Sato T, Mayanagi S, Torigoe K, Oshita A, Yamamoto H, Daiko H. Thermogenesis induced by amino acid administration prevents intraoperative hypothermia and reduces postoperative infectious complications after thoracoscopic esophagectomy. Dis Esophagus. 2017 Jan 1;30(1):1-7. doi: 10.1111/dote.12460. PMID 27003457
- [Background] Li J, Dong B, Hao D. [Clinical therapeutic effect of dexmedetomidine on patients during the extubation period of general anesthesia]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2015 Aug;40(8):898-901. doi: 10.11817/j.issn.1672-7347.2015.08.012. Chinese. PMID 26333499
- [Background] Bajwa SJ, Gupta S, Kaur J, Singh A, Parmar S. Reduction in the incidence of shivering with perioperative dexmedetomidine: A randomized prospective study. J Anaesthesiol Clin Pharmacol. 2012 Jan;28(1):86-91. doi: 10.4103/0970-9185.92452. PMID 22345953
- [Background] Ryan KF, Price JW, Warriner CB, Choi PT. Persistent hypothermia after intrathecal morphine: case report and literature review. Can J Anaesth. 2012 Apr;59(4):384-8. doi: 10.1007/s12630-011-9650-z. Epub 2011 Dec 10. PMID 22161244
- [Background] Lopez MB. Postanaesthetic shivering - from pathophysiology to prevention. Rom J Anaesth Intensive Care. 2018 Apr;25(1):73-81. doi: 10.21454/rjaic.7518.251.xum. PMID 29756066
- [Result] Seo J, Park JH, Song EH, Lee YS, Jung SK, Jeon SR, Rhim SC, Roh SW. Postoperative Nonpathologic Fever After Spinal Surgery: Incidence and Risk Factor Analysis. World Neurosurg. 2017 Jul;103:78-83. doi: 10.1016/j.wneu.2017.03.119. Epub 2017 Apr 2. PMID 28377245